CLINICAL TRIAL: NCT07211503
Title: Evaluating Correlation Ccrd Blood IL 6 and Neonatal Outcome and CTG Inflammatory Pattern
Brief Title: IL-6 and Lactates in Cord Blood and Neonatal Outcomes
Acronym: ECCO-IL6
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7963
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Fetal Infection; Fetal Inflammatory Response Syndrome; Chorioamnionitis; Chorioamnionitis Affecting Fetus or Newborn
Keywords: il6; chorioamnionitis; FIRS; lactates; labour
MeSH Terms: conditions — fetal inflammatory response syndrome; Chorioamnionitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cord blood and maternal venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SOFI group: Women with a CTG trace suspicious for fetal infection/inflammation
  Interventions: Other: blood sampling
- NEFI group: Women with normal CTG tracings and no signs of inflammation.
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — The study involves the collection of an additional aliquot of cord blood and an additional aliquot of maternal venous blood.

SUMMARY:
The goal of this observational study or clinical trial is to evaluate interleukin-6 (IL-6) and lactate levels in maternal and cord blood to identify early signs of fetal inflammation or infection.

Two groups of women with full-term pregnancies will be compared: • Case group (SOFI): women with a cardiotocograph (CTG) pattern suspicious for fetal infection/inflammation • Control group (NEFI): women with a normal cardiotocograph (CTG) pattern without signs of inflammation. The primary outcome is to evaluate whether IL-6 levels detected in the umbilical artery, alone or in combination with maternal IL-6 values, are associated with a cardiotocograph (CTG) pattern suggestive of fetal inflammation and/or a clinical picture suggestive of chorioamnionitis. Identifying a possible correlation between IL-6/lactate levels and fetal inflammatory status could facilitate more timely treatment of at-risk infants in the future, contributing to the reduction of adverse outcomes both in the neonatal period and in the long-term.

Secondary outcome are: -Comparison of fetal and maternal IL-6 levels between infants with a composite adverse outcome; - Comparison of fetal and maternal IL-6 levels in patients with and without signs of histological chorioamnionitis.

ELIGIBILITY:
Inclusion Criteria:

SOFI case group:

* Women with gestational age >37 weeks who access the delivery room of the Obstetrics and Obstetric Pathology Unit for labor.
* Single fetus in cephalic presentation
* Age ≥18 years
* Presence of CTG characteristics associated with fetal inflammation/infection (fetal heart rate (fetal heart rate (FHR) >150 bpm with gestational age >40 weeks or a 10% increase in FHR, absence of cycling, fetal tachycardia >=160 bpm, variability <5 bpm)
* Signed informed consent form by the patient.

NEFI control group:

* Women with gestation >37 weeks who access the delivery room of the Obstetrics and Obstetric Pathology Unit for labor.
* Single fetus in cephalic presentation.
* Age ≥18 years.
* Patients with a CTG tracing that does not show features associated with fetal inflammation/infection (fetal heart rate (FHR) between 110-150 bpm, normal cycling, and normal variability between 5 and 25 bpm).
* Patient signed informed consent form.

Exclusion Criteria:

* Failure to sign informed consent
* Intrauterine fetal death
* Congenital fetal and/or chromosomal abnormalities
* Maternal cardiac abnormalities and/or cardiac therapy and/or therapy with a direct effect on maternal heart rate (e.g., labetalol, digoxin)
* Twin or multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Case group - SOFI: Women in labor at term with a CTG showing criteria "Suggestive for Fetal Inflammation." Control group - NEFI: Women in labor at term with a CTG showing no inflammation/infection characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
fetal and maternal IL6 levels | 1 day
  Comparison of fetal and maternal IL-6 levels between CTGs with "Suggestive for Fetal Inflammation" (SOFI) criteria and those with "Non Evidence of Fetal Inflammation" (NEFI)

SECONDARY OUTCOMES:
IL6 and neonatal outcome | 15 days
  Comparison of fetal and maternal IL-6 levels between newborns with a composite adverse outcome
IL6 and histopathology | 1 month
  Comparison of fetal and maternal IL-6 levels in patients with and without signs of histological chorioamnionitis.

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Di Pasquo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Policlinico Gemelli, Roma, RM, Italy

REFERENCES:
- [Background] Chan CJ, Summers KL, Chan NG, Hardy DB, Richardson BS. Cytokines in umbilical cord blood and the impact of labor events in low-risk term pregnancies. Early Hum Dev. 2013 Dec;89(12):1005-10. doi: 10.1016/j.earlhumdev.2013.08.017. Epub 2013 Sep 14. PMID 24045131
- [Background] Su H, Chang SS, Han CM, Wu KY, Li MC, Huang CY, Lee CL, Wu JY, Lee CC. Inflammatory markers in cord blood or maternal serum for early detection of neonatal sepsis-a systemic review and meta-analysis. J Perinatol. 2014 Apr;34(4):268-74. doi: 10.1038/jp.2013.186. Epub 2014 Jan 23. PMID 24457256
- [Background] Kim CJ, Yoon BH, Romero R, Moon JB, Kim M, Park SS, Chi JG. Umbilical arteritis and phlebitis mark different stages of the fetal inflammatory response. Am J Obstet Gynecol. 2001 Aug;185(2):496-500. doi: 10.1067/mob.2001.116689. PMID 11518916
- [Background] Tsukimori K, Komatsu H, Yoshimura T, Hikino S, Hara T, Wake N, Nakano H. Increased inflammatory markers are associated with early periventricular leukomalacia. Dev Med Child Neurol. 2007 Aug;49(8):587-90. doi: 10.1111/j.1469-8749.2007.00587.x. PMID 17635203
- [Background] Daskalakis G, Papapanagiotou A, Siristatidis C, Drakakis P, Mole I, Barbouni A, Papavassiliou AG, Pergialiotis V. The influence of delayed cord clamping and cord milking on inflammatory cytokines in umbilical vein and neonatal circulation. Acta Obstet Gynecol Scand. 2018 May;97(5):624-628. doi: 10.1111/aogs.13294. Epub 2018 Feb 8. PMID 29338067
- [Background] Aydin I, Aydin FN, Agilli M. The evaluation of inflammatory markers in umbilical cord blood. Fetal Pediatr Pathol. 2014 Jun;33(3):196-7. doi: 10.3109/15513815.2014.898722. Epub 2014 Mar 27. PMID 24673641
- [Background] Oh JW, Park CW, Moon KC, Park JS, Jun JK. The relationship among the progression of inflammation in umbilical cord, fetal inflammatory response, early-onset neonatal sepsis, and chorioamnionitis. PLoS One. 2019 Nov 19;14(11):e0225328. doi: 10.1371/journal.pone.0225328. eCollection 2019. PMID 31743377
- [Background] Mestan K, Yu Y, Thorsen P, Skogstrand K, Matoba N, Liu X, Kumar R, Hougaard DM, Gupta M, Pearson C, Ortiz K, Bauchner H, Wang X. Cord blood biomarkers of the fetal inflammatory response. J Matern Fetal Neonatal Med. 2009 May;22(5):379-87. doi: 10.1080/14767050802609759. PMID 19529994
- [Background] Ren J, Qiang Z, Li YY, Zhang JN. Biomarkers for a histological chorioamnionitis diagnosis in pregnant women with or without group B streptococcus infection: a case-control study. BMC Pregnancy Childbirth. 2021 Mar 25;21(1):250. doi: 10.1186/s12884-021-03731-7. PMID 33765949
- [Background] Varner MW, Marshall NE, Rouse DJ, Jablonski KA, Leveno KJ, Reddy UM, Mercer BM, Iams JD, Wapner RJ, Sorokin Y, Thorp JM, Malone FD, Carpenter M, O'Sullivan MJ, Peaceman AM, Hankins GD, Dudley DJ, Caritis SN; The Eunice Kennedy Shriver National Institute of Child Health Human Development Maternal-Fetal Medicine Units Network. The association of cord serum cytokines with neurodevelopmental outcomes. Am J Perinatol. 2015 Feb;30(2):115-22. doi: 10.1055/s-0034-1376185. Epub 2014 Jun 17. PMID 24936937
- [Background] Sorokin Y, Romero R, Mele L, Iams JD, Peaceman AM, Leveno KJ, Harper M, Caritis SN, Mercer BM, Thorp JM, O'Sullivan MJ, Ramin SM, Carpenter MW, Rouse DJ, Sibai B. Umbilical cord serum interleukin-6, C-reactive protein, and myeloperoxidase concentrations at birth and association with neonatal morbidities and long-term neurodevelopmental outcomes. Am J Perinatol. 2014 Sep;31(8):717-26. doi: 10.1055/s-0033-1359723. Epub 2013 Dec 11. PMID 24338120
- [Background] Romero R, Chaemsaithong P, Docheva N, Korzeniewski SJ, Tarca AL, Bhatti G, Xu Z, Kusanovic JP, Chaiyasit N, Dong Z, Yoon BH, Hassan SS, Chaiworapongsa T, Yeo L, Kim YM. Clinical chorioamnionitis at term V: umbilical cord plasma cytokine profile in the context of a systemic maternal inflammatory response. J Perinat Med. 2016 Jan;44(1):53-76. doi: 10.1515/jpm-2015-0121. PMID 26360486
- [Background] Gotsch F, Romero R, Kusanovic JP, Mazaki-Tovi S, Pineles BL, Erez O, Espinoza J, Hassan SS. The fetal inflammatory response syndrome. Clin Obstet Gynecol. 2007 Sep;50(3):652-83. doi: 10.1097/GRF.0b013e31811ebef6. PMID 17762416
- [Background] Jung E, Romero R, Yeo L, Diaz-Primera R, Marin-Concha J, Para R, Lopez AM, Pacora P, Gomez-Lopez N, Yoon BH, Kim CJ, Berry SM, Hsu CD. The fetal inflammatory response syndrome: the origins of a concept, pathophysiology, diagnosis, and obstetrical implications. Semin Fetal Neonatal Med. 2020 Aug;25(4):101146. doi: 10.1016/j.siny.2020.101146. Epub 2020 Oct 23. PMID 33164775
- [Background] Chandraharan E, Pereira S, Ghi T, Gracia Perez-Bonfils A, Fieni S, Jia YJ, Griffiths K, Sukumaran S, Ingram C, Reeves K, Bolten M, Loser K, Carreras E, Suy A, Garcia-Ruiz I, Galli L, Zaima A. International expert consensus statement on physiological interpretation of cardiotocograph (CTG): First revision (2024). Eur J Obstet Gynecol Reprod Biol. 2024 Nov;302:346-355. doi: 10.1016/j.ejogrb.2024.09.034. Epub 2024 Oct 2. PMID 39378709
- [Background] di Pasquo E, Fieni S, Chandraharan E, Dall'Asta A, Morganelli G, Spinelli M, Bettinelli ML, Aloe R, Russo A, Galli L, Perrone S, Ghi T. Correlation between intrapartum CTG findings and interleukin-6 levels in the umbilical cord arterial blood: A prospective cohort study. Eur J Obstet Gynecol Reprod Biol. 2024 Mar;294:128-134. doi: 10.1016/j.ejogrb.2024.01.018. Epub 2024 Jan 13. PMID 38237311